CLINICAL TRIAL: NCT02219750
Title: Comparison of Switching to Premixed Insulin With Add-on Rapid-acting Insulin in Poorly Controlled Type 2 Diabetes Treated With Basal Insulin
Brief Title: Comparison of Premixed Insulin With Basal-plus Insulin in Type 2 Diabetes Patients
Acronym: COMPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sung-Chen Liu, Mackay Memorial Hospital, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13MMHISO71,13MMHISO72
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-03

CONDITIONS: Diabetes
Keywords: premix insuiln, basal-plus insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preprandial premix therapy (Active Comparator): switch twice-daily insulin Preprandial premix therapy mean that transition of advance insulin based on the basal insulin daily total dose at study entry divided into two equal dose of preprandial NovoMix 30. Patient discontinued all pre-study oral antidiabetic drug(OAD), including sulfonylureas, glinides, Thiazolidinedione(TZD) and Dipeptidyl peptidase-4(DPP-4) inhibitor but left metformin alone
  Interventions: Drug: switch twice-daily insulin
- Basal-plus insulin (Active Comparator): switch twice-daily insulin Basal-plus insulin consisted of continued previous basal insulin and add-on once-daily insulin aspart(NovoRapid) before breakfast. The starting dose of insulin aspart was 4 unit(U) before breakfast and continued under previous basal insulin dose.
  Interventions: Drug: switch twice-daily insulin

INTERVENTIONS:
Drug: switch twice-daily insulin — compare two different insuiln regimen in basal insuln base and premixed insulin.
  NovoMix 30, drug class:biphasic insulins Lantus, drug class: long-acting insuiln Levemir, durg class: long-acting insulin NovoRapid, drug class: rapid-acting insulin
  Other Names: NovoMix® 30 Penfill®, lantus®, levemir®, NovoRapid®

SUMMARY:
Comparison of efficacy and safety of different insulin regimens between basal bolus and premixed insulin in poorly controlled type 2 diabetes

DETAILED DESCRIPTION:
This is a 24-week, prospective, open-label, randomized, parallel-group study conducted in approximately 140 patients with type 2 diabetes from Mackay Memorial Hospitals and Mackay Memorial Hospital Taitung branch. After enrollment, eligible patients will be randomized in a 1:1 ratio to either Basal-plus therapy(BPT) or Preprandial premix therapy(PPT). The effectiveness of advancing insulin therapy will be assessed at baseline and at 12 and 24 weeks after initiation of study prescription. The safety will be followed during the 24-week study period. All study procedure will be conducted after obtaining informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes.(World Health Organization classification) > 20 years of age.
* Patients who have received stable doses of any OADs for at least 12 weeks prior to the screening visit.
* treatment with basal insulin plus OADs >3 months with suboptimal glycemic control (HbA1c >7%)
* FBG <130 mg/dl or FBG ≥130 mg/dl, but daily insulin dose >0.7U/kg or had history of nocturnal hypoglycemia
* Patients who are willing and able to cooperate with study and give signed informed consent.

Exclusion Criteria:

* Patients with type 1 diabetes.
* History of severe hypoglycemia or hypoglycemia unawareness within prior 6 months.
* Patients who had received any investigational insulin for more than 3 months or who have received investigational insulin treatment within 4 weeks prior to screening visit.
* Patients hypersensitive with insulin analog or its excipients.
* Patients who are currently pregnant/lactating, or who are preparing for pregnancy or lactation.
* Renal dialysis patients, patients with severe liver disease or congestive heart failure
* BMI >40kg/m2
* Excessive insulin resistance (total daily insulin dose>2.0unit/kg)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 24week duration
  To compare the change in HbA1c from baseline to endpoint for each groups at Week 24

SECONDARY OUTCOMES:
achieving goal percentage | 24weeks duration
  To compare the proportion of patients achieving HbA1c < 7% at Week 24.
plasma glucose | 24 week duration
  To compare the changes in fasting plasma glucose (FPG) and postprandial plasma glucose (PPG) at Week 24.
weight change | 24 weeks duration
  To compare the change in body weight at each visit.
incidence of hypoglcyemia | 24 weeks duration
  To evaluate the incidence of self-reported hypoglycemia episodes.
total insulin dose | 24 weeks duration
  To estimate total insulin dose.

OTHER OUTCOMES:
C peptide | 24weeks
  to compare serum C peptide between baseline and end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chen Liu, master, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memerial Hospital, Taipei, Taiwan